CLINICAL TRIAL: NCT00515021
Title: The Effects of Night-time Versus Morning Administration of Eplerenone on the Diurnal Variation of Plasminogen Activator Inhibitor-1
Brief Title: Diurnal Variation of Plasminogen Activator Inhibitor-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, James Muldowney, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 070183
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Metabolic Syndrome X
Keywords: Metabolic syndrome; Aldosterone inhibitor; Diurnal drug regimen; PAI-1 levels
MeSH Terms: conditions — Metabolic Syndrome | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daytime then nightime dosing (Experimental): Eplerenone - 50mg, by mouth, daily, in the morning x 2 weeks followed by 100mg, by mouth, daily, in the morning x 4 weeks then patients cross over to 50mg, by mouth, daily, in the evening x 2 weeks followed by 100mg, by mouth, daily, in the evening x 4 weeks.
  Interventions: Drug: Eplerenone (Morning); Drug: Eplerenone (Night-time)
- Nighttime then daytime dosing (Experimental): Eplerenone - 50mg, by mouth, daily, in the evening x 2 weeks followed by 100mg, by mouth, daily, in the evening x 4 weeks then patients cross over to 50mg, by mouth, daily, in the morning x 2 weeks followed by 100mg, by mouth, daily, in the morning x 4 weeks.
  Interventions: Drug: Eplerenone (Morning); Drug: Eplerenone (Night-time)

INTERVENTIONS:
Drug: Eplerenone (Morning) — Eplerenone - 50mg, by mouth, daily, in the morning x 2 weeks followed by 4 weeks at 100mg.
  100mg, by mouth, daily, in the morning x 4 weeks then patients cross over to 100mg, by mouth, daily, in the evening x another 4 weeks.
  Other Names: Inspra
Drug: Eplerenone (Night-time) — Eplerenone - 50mg, by mouth, daily in the evening x 2 weeks followed by 4 weeks at 100mg
  Other Names: Inspra

SUMMARY:
To determine if nighttime administration of an aldosterone antagonist would effectively lower peak plasma Plasminogen Activator Inhibitor-1 (PAI-1) levels more effectively than morning administration.

DETAILED DESCRIPTION:
Plasminogen activator inhibitor-1, a member of the serine protease inhibitor (serpin) superfamily, is the principal inhibitor to tissue-type plasminogen activator and urokinase-type plasminogen activator. Elevated plasma PAI-1 levels, an independent cardiovascular risk factor, has been shown to be a predictor of recurrent myocardial infarction (MI). Acute changes in plasma PAI-1 after MI is a predictor of mortality. PAI-1 levels are elevated in the individuals with hypertension, insulin resistance, hypertriglyceridemia, obesity, and the constellation of risk-factors known as the metabolic syndrome. PAI-1 is synthesized in the liver, vascular endothelium, vascular smooth muscle, and visceral adipose tissue. A number of factors have been shown to regulate PAI-1, including metabolic factors such as insulin, glucose, triglycerides; inflammatory cytokines such as tumor necrosis factor-α, transforming growth factor-β, interleukin-1, and more notably, components of the renin-angiotensin-aldosterone system (RAAS), namely angiotensin II and aldosterone.

PAI-1 also has a diurnal variation with a peak plasma level occurring between 8 and 9 AM that may help explain why the incidence of acute MI is highest in the morning and why thrombolysis is least effective at that time. PAI-1's diurnal variation is been shown to be directly regulated by central and peripheral circadian pacemakers in vitro, and in vivo. Our group has observed that the diurnal variation of plasma PAI-1 levels is blunted and delayed in blind individuals who's circadian mechanisms are free running (not controlled by a central circadian pacemaker) when compared to those whose circadian rhythms are entrained (controlled by a central circadian pacemaker) (unpublished data), suggesting an additional system may modulate diurnal variation of PAI-1. As plasma renin activity (PRA) and aldosterone levels peak earlier than PAI-1 levels, they may be partially responsible. Indeed, continuous infusion of candesartan eliminated diurnal variation of aortic PAI-1 message expression in Wistar-Kyoto and spontaneously hypertensive rats, while hydralazine did not.

The use of therapies to modulate plasma PAI-1 levels in human subjects have met with variable success. Low salt diet was shown to increase plasma PAI-1 levels in normotensive subjects in a manner that correlated with plasma aldosterone levels. Twice daily treatment with quinapril (40mg) lowered plasma PAI-1 levels during the expected peak time. In a second study of twice daily quinapril compared to twice daily losartan in normotensive subjects both only had a modest effect on plasma PAI-1 levels. A third study helped to explain this finding. In a crossover study, hypertensive subjects received daily spironolactone or hydrochlorothiazide (HCTZ) in a randomized fashion. Plasma PAI-1 levels were increased after HCTZ treatment, but not significantly changed from baseline with spironolactone treatment. Spironolactone treatment, however, resulted in significantly higher aldosterone levels. The correlation between plasma aldosterone and PAI-1 that was observed at baseline and with HCTZ treatment was not observed in the spironolactone arm, suggesting that the endogenous relationship between aldosterone and PAI-1 can be disrupted by mineralocorticoid receptor antagonism.

ELIGIBILITY:
Inclusion Criteria:

* Age18-65
* Metabolic Syndrome (3 or more of the following):

  1. Blood pressure 130/85 or greater
  2. Central obesity (Waist - Male > 40", Female > 35")
  3. Fasting glucose ≥ 110 mg/dl
  4. Low HDL (Male < 40 mg/dl, Female < 50 mg/dl)
  5. Elevated Triglycerides (> 150 mg/dl)

Exclusion Criteria:

* Cigarette Use
* Renal insufficiency
* Coronary Artery Disease
* Diabetes
* Blindness
* Cerebrovascular Disease
* Secondary hypertension (renal artery stenosis, pheo, etc.)
* RAAS disease (Primary Aldosteronism, etc.)
* Other chronic illness (cancer, autoimmune or liver disease)
* Pregnancy
* Anemia (Hgb < 12 mg/dl)
* Evening or Night Shift work
* Transmeridian travel in previous 6 months
* History of sleep disorders
* Hypokalemia (serum potassium < 3.5 milliequivalent (mEq/L)
* Hyperkalemia (serum potassium > 5.5 mEq/L
* Reported hypersensitivity to HCTZ or eplerenone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Muldowney, III, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant withdrew prior to randomization
Groups:
- Eplerenone: Morning Administration Then Evening: Eplerenone - 50mg, by mouth, daily, in the morning for 2 weeks followed by 100mg, by mouth, daily, in the morning x 4 weeks
  Eplerenone - 50mg, by mouth, daily in the evening x 2 weeks followed by 4 weeks at 100mg
- Eplerenone: Evening Administration Then Morning: Eplerenone 50mg, by mouth, daily, in the evening for 2 weeks followed by 100mg, by mouth, daily, in the evening x 4 weeks
  Eplerenone - 50mg, by mouth, daily, in the morning for 2 weeks followed by 100mg, by mouth, daily, in the morning x 4 weeks
Period: Overall Study
Arm/Group | Eplerenone: Morning Administration Then Evening | Eplerenone: Evening Administration Then Morning
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eplerenone: Morning Administration Then Evening | Eplerenone: Evening Administration Then Morning | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Plasminogen Activator Inhibitor-1 (PAI-1) Levels
Description: baseline PAI-1 levels prior to drug administration
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Eplerenone: Morning Administration Then Evening | Eplerenone: Evening Administration Then Morning
Number analyzed (Participants) | 9 | 11
ng/ml | 41.5 (17.9) | 42.9 (10.5)

2. Primary Outcome: Plasminogen Activator Inhibitor-1 (PAI-1) Levels
Description: PAI-1 levels after Eplerenone 50mg daily for 2 weeks then 100mg daily for 4 weeks. Time of administration varied in the arms, either morning or night time dosing.
Time Frame: after 6 weeks on Eplerenone
Measure: Mean (Standard Error); unit: ng/ml
Groups:
- Eplerenone: Morning Administration: Eplerenone - 50mg, by mouth, daily, in the morning for 2 weeks followed by 100mg, by mouth, daily, in the morning x 4 weeks
- Eplerenone: Night-time Administration: Eplerenone 50mg, by mouth, daily, in the evening for 2 weeks followed by 100mg, by mouth, daily, in the evening x 4 weeks
Arm/Group | Eplerenone: Morning Administration | Eplerenone: Night-time Administration
Number analyzed (Participants) | 20 | 20
ng/ml | 39.9 (4.0) | 40.4 (3.8)

ADVERSE EVENTS:
Arm/Group | Eplerenone: Morning Administration Then Evening | Eplerenone: Evening Administration Then Morning
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/9 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No